CLINICAL TRIAL: NCT04192916
Title: Use of Direct Oral Anticoagulants (DOACs) in Patients With Ph-negative Myeloproliferative Neoplasms
Acronym: MPN-DOACs
Status: Completed | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: MPN-DOACs
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Myeloproliferative Neoplasm
Keywords: Efficacy and safety profile; Direct oral anticoagulants; Real world data
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Dabigatran; edoxaban; Rivaroxaban; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MPN patients treated with DOACs
  Interventions: Drug: DOACs

INTERVENTIONS:
Drug: DOACs — Direct Oral Anticoagulants
  Other Names: Dabigatran; Edoxaban; Rivaroxaban; Apixaban

SUMMARY:
Patients with myeloproliferative neoplasms (MPN) are predisposed to have an increased thrombotic and hemorrhagic risk and, in this context, the use of newly approved direct oral anticoagulants (DOACs) may have improved bleeding risk compared to warfarin use. However, the published experience is very limited and does not allow any conclusion. In the cohort of patients with MPN and venous thromboembolism (VTE) of European Leukemia-net, only 3.3% of patients had been treated with DOACs. Similarly, in a recent publication of a series of 760 patients with single-center MPN, only 25 (3.3%) were treated with a DOAC (13 for atrial fibrillation and 12 for thrombotic events).

While it is known that the risk of thrombotic recurrence and haemorrhagic event during warfarin treatment is about 30% at 5 years from the first event, the actual risk of such events in MPN patients is not known.

The aim of the present study is therefore to obtain information on patients with MPN treated with DOAC for atrial fibrillation (AF) and VTE. This is an international multi-center retrospective survey aimed at describing the efficacy / safety of DOAC in the prevention of:

* cardioembolic stroke in patients with MPN with AF
* recurrent thrombosis in patients with MPN with VTE
* major bleeding in all patients with MPN.

The results will allow to design future prospective studies that evaluate the benefit / risk profile of DOAC compared to warfarin in these pathologies characterized by high risk of thrombosis and, in some subgroups, of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Philadelphia-negative MPN according to World Health Organization (WHO) 2008 and/or 2016 criteria until 31/12/2018;
* diagnosis of atrial fibrillation (AF) and/or diagnosis of venous thromboembolism (VTE) including thrombosis of deep veins of the limbs and the abdomen, cerebral and splanchnic veins (hepatic, portal, mesenteric, and splenic veins) and pulmonary embolism;
* treatment with DOACs.

Exclusion Criteria:

• Administration of DOAC for any medical reason other than AF and/or VTE (excluding superficial vein thrombosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MPN treated with any DOAC for AF or VTE
Sampling Method: Non-Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of major thrombosis and bleeding | At 5 year from the start of treatment with DOACs
  Cumulative incidence of major arterial and venous thrombosis and major bleeding as defined by the International Society on Thrombosis and Haemostasis (ISTH)

CONTACTS AND LOCATIONS:
Locations (18):
- Mount Sinai New York, New York, New York, United States
- Princess Margaret Cancer Centre Toronto, Toronto, Canada
- Centre Hospitalier Universitaire de Brest, Brest, France
- Germany (2):
  - RWTH Aachen University, Aachen
  - Johannes Wesling Klinikum Minden, Minden
- Italy (11):
  - Divisione Ematologia, Ospedale Borgo Roma, Verona, Veneto
  - ASST- Papa Giovanni XXIII - S.I.M.T., Bergamo
  - Policlinico S. Orsola - Malpighi, Bologna
  - AOU Careggi di Firenze, Florence
  - ASST MONZA Ospedale San Gerardo Clinica Ematologica, Monza
  - Azienda Ospedaliera Universitaria Federico II di Napoli Divisione di Ematologia e Trapianti del Midollo, Napoli
  - AOU Policlinico di Palermo, Palermo
  - Fondazione IRCCS Policlinico San Matteo S.C Ematologia, Pavia
  - Fondazione Policlinico Universitario A. Gemelli IRCCS UCSC Ematologia, Roma
  - A.O.U. Città della Salute e della Scienza di Torino - Ospedale Molinette- S.C. Ematologia, Torino
  - Ospedale San Bortolo di Vicenza - U.O.C di Ematologia, Vicenza
- Hospital Clinic, Hematology Department, Barcelona, Spain
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided